CLINICAL TRIAL: NCT06051513
Title: Colistimethate Sodium for Injection in The Treatment of Carbapenem-Resistant Enterobacteriaceae Infection：a Prospective, Open-label, Randomized Controlled, Multicenter Clinical Trial
Brief Title: Efficacy and Safety of Colistimethate Sodium for Injection in The Treatment of Carbapenem-Resistant Enterobacteriaceae Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Principal Investigator, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COUNT-CRE
Record Dates: First submitted 2023-09-07; First posted 2023-09-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection
Keywords: Colistimethate Sodium for Injection; Hospital-acquired pneumonia; Bloodstream infection; Carbapenem-resistant Enterobacteriaceae
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Sepsis | interventions — Therapeutics; Colistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colistin group (Experimental): For patients in this group, colistin based therapy is used. Colistin combined with metroperan or imipenem（MIC≤8mg/L），or colistin combined with tigecycline, or colistin combined with aminoglycosides (amikacin) are suggested to treat patients diagnosed with hospital-acquired pneumonia or bloodstream infection caused by carbapenem-resistant enterobacteriaceae.
  At the beginning of the intravenous use of Colistimethate Sodium for Injection，the load dose is 300mg CBA(about 9 million U)，and after 12-24 hours，the first maintenance dose should be given. The daily maintenance dose was 300-360mg CBA(9 million-10.9 million U), divided into two times (1/12h), for each time, 0.5-1 hour is needed to complete the infusion.
  Drug: colistin, other name: Colistimethate Sodium for Injection
  Interventions: Drug: treatment with or without colistin
- control group (Active Comparator): For patients in this group,best available treatment without colistin is used. Ceftazidime-avibactam, tigecycline combined with metroperan or imipenem（MIC≤8mg/L）, tigecycline combined with aminoglycosides (amikacin) are suggested to treat patients diagnosed with hospital-acquired pneumonia or bloodstream infection caused by carbapenem-resistant enterobacteriaceae.Dose of other drugs are listed below: 1-2g meropenem should be given every 8 hours，1g Imipenem every 8 hours or 6 hours，0.8g Amikacin everyday，2.5g ceftazidime-avibactam every 8 hours. A load dose of 200mg tigecycline is needed, followed by 100mg every 12 hours.
  Interventions: Drug: treatment with or without colistin

INTERVENTIONS:
Drug: treatment with or without colistin — For patients in this treatment group, colistin based therapy is used. Colistin combined with metroperan or imipenem（MIC≤8mg/L），or colistin combined with tigecycline, or colistin combined with aminoglycosides (amikacin) are suggested to treat patients diagnosed with hospital-acquired pneumonia or bloodstream infection caused by carbapenem-resistant enterobacteriaceae. For patients in the control, best available treatment without colistin is uesed; Ceftazidime-avibactam, tigecycline combined with metroperan or imipenem（MIC≤8mg/L）, tigecycline combined with aminoglycosides (amikacin) are suggested to treat patients diagnosed with hospital-acquired pneumonia or bloodstream infection caused by carbapenem-resistant enterobacteriaceae.

SUMMARY:
Colistin can be used to treat the infection caused by carbapenem-resistant enterobacteriaceae(CRE). In China, patients diagnosed with Hospital-acquired-pneumonia (HAP)or bloodstream infection caused by CRE are recruited, and randomly assigned to two groups, and in one group the patients accept treatment with colistin, however in another group, the patients accept treatment without colistin. The efficacy and safety of the treatment between the two groups are compared.

DETAILED DESCRIPTION:
The study will be conducted in accordance with good clinical practice and with the guidelines set out in the Declaration of Helsinki. After approval from local and national ethics committees, patients diagnosed with Hospital-acquired-pneumonia (HAP)or bloodstream infection caused by CRE from 14 centres in China will be recruited. All patients will be randomized to receive treatment with or without colistin in the ICU. The purpose of this study is to investigate the efficacy and safety of colistin when used to treat patients with CRE infection. The primary outcome is 14-day all cause mortality and the second outcomes include 14-day clinical cure rate, 14-day efficacy rate, ICU free days within 28 days after randomization，14-day microbiological cure rate，incidence of adverse events and severe adverse events in first 14 days, hospital mortality, 28-day all cause mortality, ICU mortality. Clopper-Pearson method is used to calculate the 95% confidence interval of mortality, Miettinen and Nurminen method is used to detect the difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who can provide written informed consent or their informed consent can be provided by legal guardian
2. Patients who are hospitalized
3. Adults ≥18 years and ≤85 years of age
4. Patients suspected of or diagnosed with hospital-acquired pneumonia (HAP, in a patient hospitalised for more than 48 hours or developing within 7 days after discharge from a hospital) or bloodstream infection caused carbapenem-resistant enterobacteriaceae (CRE) based on the culture results of the sample collected 5 days before the randomization or rapid diagnostic detection.

   Rapid testing of respiratory or blood specimens should be used to enable early identification of CRE infection pneumonia. Patients can be randomized based on the results of the rapid test while awaiting results of cultures from the local laboratory. However, if the sample does not grow CRE in the local microbiology laboratory culture, these patients will be withdrawn from the study drug treatment.

   Patients with HAP should fulfil one of the following systemic signs: 1)Fever (temperature >38°C) or hypothermia (rectal/core temperature <35°C);2)White blood cell (WBC) count >10,000 cells/mm3, or WBC count <4500 cells/mm3, or >15% band forms and fulfil at least two of the following respiratory signs or symptoms:1)a new onset of cough (or worsening of cough);2)production of purulent sputum or endotracheal secretions;3)auscultatory findings consistent with pneumonia/pulmonary consolidation (e.g., rales, rhonchi, bronchial breath sounds, dullness to percussion, egophony);4)dyspnoea, tachypnoea or hypoxaemia (O2 saturation <90% or pO2 <60 mmHg while breathing room air).

   Patients with bloodstream infection should fulfil one of the following criterion:1)fever(≥38 ℃);2)chills;3)hypotension(systolic <90 mmHg, requiring vasopressors to maintain mean arterial pressure ≥60 mmHg,decreased by 30mmHg from baseline) ,and isolation of CRE from at least two blood culture collected from two different sites.
5. Respiratory or blood specimen obtained for culture within 5 days prior to randomization, and after the onset of signs and symptoms of HAP or bloodstream infection (ideally before receipt of any systemic antibiotics).
6. Patients whose APACHE II score is between 10 and 30.

Exclusion Criteria:

1. Patients who received polymyxin for more than 48 hours in the 72 hours prior to randomization.
2. Patients who received antibiotics more than 24 hours in the 72 hours prior to randomization, and after treatment，conditions of patients improved.
3. Patient with history of serious allergy, hypersensitivity (eg, anaphylaxis), or any serious reaction to Colistimethate Sodium for Injection or other ingredients of it.
4. Evidence of active concurrent pneumonia requiring additional antimicrobials treatment caused by Streptococcus pneumoniae，Haemophilus influenzae，Methicillin-resistant staphylococcus aureus，Vancomycin-resistant enterococcus，Mycoplasma pneumonia，Legionella pneumophila, respiratory syncytial virus, influenza virus, parainfluenza virus, Middle East Respiratory Virus, Mycobacteria, Aspergillus, Mucormycosis, Candida,etc. If these organisms are identified but it is deemed by the Investigator that no treatment is warranted and their presence does not significantly change the prognosis of the patient, then the patient may be considered for this study.
5. Patients who are diagnosed with primary lung cancer (including small cell lung cancer/non-small cell lung cancer patients) or other malignancy transferred to the lungs or other known post obstructive pneumonia. Patients who is known or suspected of active tuberculosis, cystic fibrosis, lung abscess, pyothorax or obstructive pneumonia.
6. Patients with hematological malignancy such as leukemia, lymphoma and multiple myeloma.
7. Patients with lung/heart transplantation or stem cell transplantation.
8. Patient was immunocompromised and at risk of infection by opportunistic pathogens including, but not limited to the following:1) HIV (AIDS or CD4 <200). 2) chemoradiotherapy within 3 months prior to randomisation. 3) Immunosuppressive therapy including maintenance corticosteroids (0.5 mg/kg prednisone per day or other equivalent glucocorticoid). 4) Absolute neutrophil count <500/mm3.
9. Patients with chronic liver failure with portal hypertension, acute hepatic failure or acute decompensation of chronic hepatic failure.
10. Patients who participated in other clinical trials within three months.
11. Patient was pregnant or breastfeeding. If either urine or serum β-hCG test was positive, the patient was excluded.
12. Patient who have been previously enrolled in this study.
13. Patients who have condionts that may affect the trial.
14. Other conditions exist researchers thought are not suitable.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
14-day all cause mortality | from randomization to day 14
  the proportion of subjects who die within 14 days after randomization to the number of subjects in each group

SECONDARY OUTCOMES:
14-day clinical cure rate | from randomization to day 14
  the proportion of subjects who are thought as clinical effectiveness 14 days after randomization to the number of subjects in each group.
14-day efficacy rate | from randomization to day 14
  the proportion of subjects of who are thought as recovery 14 days after randomization to the number of subjects in each group.
ICU free days within 28 days after randomization | from randomization to day 28
  days that patients are not treated in ICU within 28 days after randomization of each patient in each group. If the patient die within 28 days, it will be zero.
14-day microbiological cure rate | from randomization to day 14
  the proportion of subjects of microbiological cure to the number of subjects in each group 14 days after randomization.
incidence of adverse events and severe adverse events within first 28 days | from randomization to day 28
  the proportion of patients who experience adverse events and severe adverse events within 14 days after randomization to the number of subjects in each group wihtin first 14 days
hospital mortality | to be evaluated up to 90 days post randomization
  the proportion of subjects who die when treated in hospital to the number of subjects in each group
28-day all cause mortality | from randomization to day 28
  the proportion of subjects who die within 28 days after randomization to the number of subjects in each group
ICU mortality | to be evaluated up to 90 days post randomization
  the proportion of subjects who die in ICU to the number of subjects in each group

CONTACTS AND LOCATIONS:
Overall Officials: Yingzi Huang, MD, Study Chair — Department of Critical Care Medicine, Zhongda Hospital, School of Medicine, Southeast University
Locations (15):
- China (15):
  - Anhui Provincial People's Hospital, Hefei, Anhui
  - The First Hospital of Anhui Medical University, Hefei, Anhui
  - Jinjiang Municipal Hospitall, Jinjiang, Fujian
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - The First Hospital of Lianyungang, Lianyungang, Jiangsu
  - Zhongda Hospital Affiliated to Southeast University, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Suzhou Municipal Hospitial, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - JiangsuTaizhou People's Hospital, Taizhou, Jiangsu
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Yancheng No.1 People's Hospital, Yancheng, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Yixing People's Hospital, Yixing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Zhang C, Li J, Chen T, Xie J, Huang Y. Multicentre open-label randomised controlled trial comparing the efficacy and safety of colistin-based combination therapy with the best available therapy for treating hospital-acquired pneumonia or bloodstream infections caused by carbapenem-resistant Enterobacteriaceae (COUNT-CRE): a study protocol. BMJ Open. 2025 Jul 16;15(7):e092157. doi: 10.1136/bmjopen-2024-092157. PMID 40669898